CLINICAL TRIAL: NCT06534931
Title: Effects of a High Velocity Low Amplitude Mid-Thoracic Spinal Segment Manipulation on the Force Output of the Hip Adductors and Extensors and the Latissimus Dorsi in Healthy Individuals With Unilateral Hip Adductor Weakness
Brief Title: Effects of a Thoracic Manipulation on Hip Adductor, Extensor, and Latissimus Dorsi Force in Those With Adductor Weakness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Collaborators: Raymond Chiropractic (Unknown)
Responsible Party: Principal Investigator, Michael Lawrence, Associate Teaching Professor, University of New England
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ThoracicManip
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were unaware of the existence of a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manipulation (Experimental): Those in the intervention group received a high velocity low amplitude manipulation to the mid-thoracic spine provided by a licensed chiropractor.
  Interventions: Procedure: High velocity low amplitude thoracic spine manipulation
- Sham (Sham Comparator): Those in the control group received a validated sham manipulation to the mid-thoracic spine. The sham manipulation was done so that there was minimal downward force applied to the spine.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: High velocity low amplitude thoracic spine manipulation — Participants were supine on a treatment table. The chiropractor determined levels of apparent spinal dysfunction by means of static palpation. Participants were then asked to curl forward and bring their knees to their chest as the chiropractor placed a fist just inferior to the targeted level, anywhere between the T4 - T10 vertebrae. The participant was instructed to inhale and then exhale, at which point the chiropractor lowered the participant's torso back to the table and delivered a thrust using his body into his fist.
  Arms: Manipulation
Procedure: Sham — A previously validated physiologically inert manual procedure to the thoracic spine
  Arms: Sham

SUMMARY:
The goal of this trial was to determine if a mid-thoracic high velocity low amplitude spinal manipulation improves force output in those with unilateral hip adductor weakness. The main aims were to determine if the intervention:

Improved hip adductor force and muscle activation immediately and 48 h post manipulation compared to a control group.

Improved gluteus maximus and latissimus dorsi force and muscle activation immediately and 48 h post manipulation compared to a control group.

Strength and muscle activation of the hip adductors, hip extensors (gluteus maximus), and shoulder extensors (latissimus dorsi) were measured prior to, immediate after, and 48 hours after receiving a high velocity low amplitude manipulation to the thoracic spine. The manipulation was performed by a licensed chiropractor.

A control group received a validated sham manipulation to the thoracic spine. Participants were blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hip adductor weakness, as assessed by manual muscle testing
* Pain free hip motion
* No contraindications to high velocity thoracic spine manipulation including:

Any known active cancer/ Metastatic Bone Cancer Osteoporosis or other metabolic bone disorders Signs of spinal cord compression Nerve root compression with increasing neurologic deficit Signs of Vertebrobasilar insufficiency/ cervical artery abnormalities Bleeding Diatheses Angina pectoris

Exclusion Criteria:

* Current pain in the adductor muscle group
* Past history of hip surgery
* Past history of hip fracture
* History of spine or rib fractures
* Psoas muscle group (hip flexor) weakness as determined by manual muscle testing
* Received a chiropractic manipulation in past week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Hip adductor force (weak limb) | Pre intervention, immediatly post intervention, 48 hours post intervention
  Isometric force produced by the hip adductors in the weaker limb. Measured with a force transducer and reported in Newtons.
Hip adductor muscle activity (weak limb) | Pre intervention, immediatly post intervention
  Mean muscle activity during isometric contraction. Measured with surface electrode and reported as a percentage of maximum activation.

SECONDARY OUTCOMES:
Hip extension force (strong limb) | Pre intervention, immediatly post intervention, 48 hours post intervention
  Isometric force produced by the hip extensors in the strong limb. Measured with a force transducer and reported in Newtons.
Gluteus maximus muscle activity (strong limb) | Pre intervention, immediatly post intervention
  Mean muscle activity during isometric contraction. Measured with surface electrode and reported as a percentage of maximum activation.
Hip extension force (weak limb) | Pre intervention, immediatly post intervention, 48 hours post intervention
  Isometric force produced by the hip extensors in the weak limb. Measured with a force transducer and reported in Newtons.
Gluteus maximus muscle activity (weak limb) | Pre intervention, immediatly post intervention
  Mean muscle activity during isometric contraction. Measured with surface electrode and reported as a percentage of maximum activation.
Shoulder extension force (weak limb) | Pre intervention, immediatly post intervention, 48 hours post intervention
  Isometric force produced by the shoulder extensors in the weak limb. Measured with a force transducer and reported in Newtons.
Latissimus dorsi muscle activity (weak limb) | Pre intervention, immediatly post intervention
  Mean muscle activity during isometric contraction. Measured with surface electrode and reported as a percentage of maximum activation.
Shoulder extension force (strong limb) | Pre intervention, immediatly post intervention, 48 hours post intervention
  Isometric force produced by the shoulder extensors in the strong limb. Measured with a force transducer and reported in Newtons.
Latissimus dorsi muscle activity (strong limb) | Pre intervention, immediatly post intervention
  Mean muscle activity during isometric contraction. Measured with surface electrode and reported as a percentage of maximum activation.
Hip adductor muscle activity (strong limb) | Pre intervention, immediatly post intervention
  Mean muscle activity during isometric contraction. Measured with a force transducer and reported in Newtons.
Hip adductor force (strong limb) | Pre intervention, immediatly post intervention, 48 hours post intervention
  Isometric force produced by the hip adductors in the strong limb. Measured with a force transducer and reported in Newtons.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New England, Portland, Maine, United States

REFERENCES:
- [Background] Haavik H, Kumari N, Holt K, Niazi IK, Amjad I, Pujari AN, Turker KS, Murphy B. The contemporary model of vertebral column joint dysfunction and impact of high-velocity, low-amplitude controlled vertebral thrusts on neuromuscular function. Eur J Appl Physiol. 2021 Oct;121(10):2675-2720. doi: 10.1007/s00421-021-04727-z. Epub 2021 Jun 23. PMID 34164712
- [Background] Christiansen TL, Niazi IK, Holt K, Nedergaard RW, Duehr J, Allen K, Marshall P, Turker KS, Hartvigsen J, Haavik H. The effects of a single session of spinal manipulation on strength and cortical drive in athletes. Eur J Appl Physiol. 2018 Apr;118(4):737-749. doi: 10.1007/s00421-018-3799-x. Epub 2018 Jan 11. PMID 29327170
- [Background] Holt K, Niazi IK, Nedergaard RW, Duehr J, Amjad I, Shafique M, Anwar MN, Ndetan H, Turker KS, Haavik H. The effects of a single session of chiropractic care on strength, cortical drive, and spinal excitability in stroke patients. Sci Rep. 2019 Feb 25;9(1):2673. doi: 10.1038/s41598-019-39577-5. PMID 30804399
- [Background] Niazi IK, Kamavuako EN, Holt K, Janjua TAM, Kumari N, Amjad I, Haavik H. The Effect of Spinal Manipulation on the Electrophysiological and Metabolic Properties of the Tibialis Anterior Muscle. Healthcare (Basel). 2020 Dec 10;8(4):548. doi: 10.3390/healthcare8040548. PMID 33321904
- [Background] Niazi IK, Turker KS, Flavel S, Kinget M, Duehr J, Haavik H. Changes in H-reflex and V-waves following spinal manipulation. Exp Brain Res. 2015 Apr;233(4):1165-73. doi: 10.1007/s00221-014-4193-5. Epub 2015 Jan 13. PMID 25579661
- [Background] Chilibeck PD, Cornish SM, Schulte A, Jantz N, Magnus CR, Schwanbeck S, Juurlink BH. The effect of spinal manipulation on imbalances in leg strength. J Can Chiropr Assoc. 2011 Sep;55(3):183-92. PMID 21886280
- [Background] Grindstaff TL, Hertel J, Beazell JR, Magrum EM, Ingersoll CD. Effects of lumbopelvic joint manipulation on quadriceps activation and strength in healthy individuals. Man Ther. 2009 Aug;14(4):415-20. doi: 10.1016/j.math.2008.06.005. Epub 2008 Sep 20. PMID 18805726
- [Background] Hillermann B, Gomes AN, Korporaal C, Jackson D. A pilot study comparing the effects of spinal manipulative therapy with those of extra-spinal manipulative therapy on quadriceps muscle strength. J Manipulative Physiol Ther. 2006 Feb;29(2):145-9. doi: 10.1016/j.jmpt.2005.12.003. PMID 16461174
- [Background] Botelho MB, Andrade BB. Effect of cervical spine manipulative therapy on judo athletes' grip strength. J Manipulative Physiol Ther. 2012 Jan;35(1):38-44. doi: 10.1016/j.jmpt.2011.09.005. Epub 2011 Nov 10. PMID 22079053
- [Background] Fernandez-Carnero J, Fernandez-de-las-Penas C, Cleland JA. Immediate hypoalgesic and motor effects after a single cervical spine manipulation in subjects with lateral epicondylalgia. J Manipulative Physiol Ther. 2008 Nov-Dec;31(9):675-81. doi: 10.1016/j.jmpt.2008.10.005. PMID 19028251
- [Background] Dishman JD, Ball KA, Burke J. First Prize: Central motor excitability changes after spinal manipulation: a transcranial magnetic stimulation study. J Manipulative Physiol Ther. 2002 Jan;25(1):1-9. PMID 11898013
- [Background] Hegedus EJ, Goode A, Butler RJ, Slaven E. The neurophysiological effects of a single session of spinal joint mobilization: does the effect last? J Man Manip Ther. 2011 Aug;19(3):143-51. doi: 10.1179/2042618611Y.0000000003. PMID 22851877
- [Background] Lawrence MA, Raymond JT, Look AE, Woodard NM, Schicker CM, Swanson BT. Effects of Tibiofibular and Ankle Joint Manipulation on Hip Strength and Muscle Activation. J Manipulative Physiol Ther. 2020 Jun;43(5):406-417. doi: 10.1016/j.jmpt.2019.10.005. Epub 2020 Jul 20. PMID 32703611
- [Background] Michener LA, Kardouni JR, Lopes Albers AD, Ely JM. Development of a sham comparator for thoracic spinal manipulative therapy for use with shoulder disorders. Man Ther. 2013 Feb;18(1):60-4. doi: 10.1016/j.math.2012.07.003. Epub 2012 Aug 9. PMID 22883130
- [Background] Parkinson AO, Apps CL, Morris JG, Barnett CT, Lewis MGC. The Calculation, Thresholds and Reporting of Inter-Limb Strength Asymmetry: A Systematic Review. J Sports Sci Med. 2021 Oct 1;20(4):594-617. doi: 10.52082/jssm.2021.594. eCollection 2021 Dec. PMID 35321131